CLINICAL TRIAL: NCT05860179
Title: Analyzing Factors of Patient Involvement in Multiple Myeloma Clinical Trials
Brief Title: Examination of Trends in Multiple Myeloma Trial Patient Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80736578
Record Dates: First submitted 2023-04-21; First posted 2023-05-16 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical trials has been highly skewed towards specific demographic groups. However, research identifying which trial attributes impact participation, in either positive or negative ways, is limited.

This study invites participants to record a wide range of data on their clinical trial experience, with the goal being to identify factors which persistently limit patients' ability to participate in, or complete, a trial in which they were initially interested.

Data will be analyzed through a range of demographic lenses, in hopes of discovering patterns which might improve the experience of future multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patient has been diagnosed with multiple myeloma
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form
* Pregnant, breastfeeding or expecting to conceive within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple myeloma patients who are actively considering enrolling in a medical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with multiple myeloma who decide to enroll in clinical trial | 3 Months
Rate of patients with multiple myeloma who remain in clinical trial to completion | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes LL, Zhou J, Kanapuru B, Horodniceanu E, Gwise T, Kluetz PG, Bhatnagar V. Review of patient-reported outcomes in multiple myeloma registrational trials: highlighting areas for improvement. Blood Cancer J. 2021 Aug 31;11(8):148. doi: 10.1038/s41408-021-00543-y. PMID 34465728
- [Background] Goldschmidt H. [Clinical update-multiple myeloma]. Radiologe. 2022 Jan;62(1):3-11. doi: 10.1007/s00117-021-00941-0. Epub 2021 Dec 30. German. PMID 34967910
- [Background] Efficace F, Cottone F, Sparano F, Caocci G, Vignetti M, Chakraborty R. Patient-Reported Outcomes in Randomized Controlled Trials of Patients with Multiple Myeloma: A Systematic Literature Review of Studies Published Between 2014 and 2021. Clin Lymphoma Myeloma Leuk. 2022 Jul;22(7):442-459. doi: 10.1016/j.clml.2022.01.009. Epub 2022 Jan 19. PMID 35183476

DOCUMENTS (1):
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05860179/ICF_000.pdf